CLINICAL TRIAL: NCT07381257
Title: Efficacy and Safety of Rifaximin-α in the Treatment of Metabolic Dysfunction-Associated Steatotic Liver Disease: A Randomized, Open-Label, Controlled Pilot Clinical Trial
Brief Title: Efficacy and Safety of Rifaximin-α in Treating MASLD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZXH2025010.10
Record Dates: First submitted 2025-12-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Metabolic Dysfunction-Associated Steatotic Liver Disease; Rifaximin

STUDY DESIGN:
Intervention Model Description: Enrolled MASLD patients will be randomized in a 2:1 ratio to the rifaximin-α treatment group (40 cases) or the control group (20 cases). All patients are advised to maintain daily physical activity and follow a recommended dietary plan (e.g., Mediterranean diet). The Rifaximin treatment group will receive oral Rifaximin-α at a dose of 1200 mg per day for 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients are advised to maintain daily physical activity and follow a recommended dietary plan (e.g., Mediterranean diet).
- Treatmnet group (Experimental): The Rifaximin treatment group will receive oral Rifaximin-α at a dose of 1200 mg per day for 24 weeks. And patients are advised to maintain daily physical activity and follow a recommended dietary plan (e.g., Mediterranean diet).
  Interventions: Drug: Rifaximin-α (Alfa Wassermann S.p.A., Italy)

INTERVENTIONS:
Drug: Rifaximin-α (Alfa Wassermann S.p.A., Italy) — Participants in the treatment group will receive oral Rifaximin-α at a dosage of 1200 mg/day (400 mg, three times daily) for 24 weeks.
  Arms: Treatmnet group

SUMMARY:
Study Objective: To evaluate the efficacy and safety of Rifaximin-α in the treatment of Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD), and investigate the underlying mechanisms by which Rifaximin-α influences MASLD progression.

Target Population: Patients diagnosed with MASLD. Intervention: This trial is a multicenter, prospective, randomized, controlled study. Enrolled MASLD patients who meet the inclusion criteria, do not meet any exclusion criteria, and provide written informed consent will be randomized in a 2:1 ratio to the Rifaximin-α treatment group (40 cases) or the control group (20 cases). All patients are advised to maintain daily physical activity and follow a recommended dietary plan (e.g., Mediterranean diet). The Rifaximin-α treatment group will receive oral Rifaximin-α at a dose of 1200 mg per day for 24 weeks. Both groups of patients will enter a 24-week follow-up period after completing the 24-week treatment. During the study, patients' existing foundational treatments (such as liver-protecting, lipid-lowering, glucose-lowering, and antihypertensive therapies) will be maintained. Relevant indicators will be closely monitored. And avoid the use of medications known to alter the gut microbiota, such as lactulose, antibiotics, and various types of intestinal microecological preparations.

Investigational Drug: Rifaximin-α (Alfa Wassermann S.p.A., Italy).

ELIGIBILITY:
Inclusion Criteria

1. Willingness to provide written informed consent.
2. Aged 18 to 75 years, inclusive, regardless of gender.
3. Diagnosis of hepatic steatosis (fatty liver) within the past 6 months.
4. Presence of at least one metabolic/cardiovascular risk factor:

   A. BMI ≥ 23.0 kg/m², or waist circumference ≥ 90 cm (male) / 80 cm (female). B. Fasting plasma glucose (FPG) ≥ 5.6 mmol/L, or 2-hour postprandial glucose ≥ 7.8 mmol/L, or HbA1c ≥ 5.7%, or documented history of type 2 diabetes mellitus (T2DM) or current use of anti-diabetic medication.

   C. Fasting serum triglycerides (TG) ≥ 1.70 mmol/L, or current use of medication for hypertriglyceridemia.

   D. Serum high-density lipoprotein (HDL) cholesterol ≤ 1.0 mmol/L (male) and ≤ 1.3 mmol/L (female), or current use of lipid-lowering medication.

   E. Blood pressure ≥ 130/85 mmHg, or current use of antihypertensive medication.
5. Liver fat content ≥ 8% as measured by Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF).

Exclusion Criteria

1. Confirmed diagnosis of liver cirrhosis based on clinical, laboratory, imaging, and/or liver biopsy findings.
2. Evidence of other specific etiologies of chronic liver disease confirmed by history or laboratory tests, including but not limited to: viral hepatitis (B or C, etc.), autoimmune liver disease, alcohol-related liver disease (defined as >20 g/day for females or >30 g/day for males), drug-induced liver injury, Wilson's disease, alpha-1 antitrypsin deficiency, or hereditary hemochromatosis.
3. Other identifiable causes of hepatic steatosis confirmed by history or laboratory tests, such as: specific medications (e.g., tamoxifen, amiodarone, valproate, methotrexate, glucocorticoids, olanzapine), total parenteral nutrition, hypothyroidism, inflammatory bowel disease, Cushing's syndrome, celiac disease, abetalipoproteinemia, lipodystrophic diabetes, Mauriac syndrome, hypopituitarism, hypogonadism, polycystic ovary syndrome, etc.
4. Use of medications known to alter gut microbiota (e.g., lactulose, systemic antibiotics, any intestinal microecological preparations) within 4 weeks prior to screening.
5. Dose of hepatoprotective or lipid-lowering medications not stabilized for at least 4 weeks prior to screening.
6. Received any Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) or remeglutide treatment within 12 weeks prior to screening, or plans to receive such treatment during the study.
7. Dose of medications that may affect MASLD, anti-diabetic agents (excluding GLP-1 RAs and remeglutide), or weight-loss drugs not stabilized for at least 12 weeks prior to screening.
8. Self-reported weight change >5% within 4 weeks prior to screening.
9. BMI > 35 kg/m².
10. Poorly controlled glycemia: HbA1c > 9%.
11. Total bilirubin > 1.5 mg/dL (except with normal direct bilirubin), or Alanine Aminotransferase (ALT) > 5 times the Upper Limit of Normal (ULN), or Aspartate Aminotransferase (AST) > 5 times ULN, or Alkaline Phosphatase (ALP) > 2 times ULN.
12. Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m².
13. History of or planned bariatric/metabolic therapy, including but not limited to endoscopic interventions, surgical procedures, or Traditional Chinese Medicine therapies. Exceptions may be made if previous interventions have been reversed or removed (e.g., intragastric balloon, subcutaneous threads) for more than 12 weeks.
14. History of or current hepatocellular carcinoma (HCC).
15. Diagnosis of any malignancy within the past 5 years, except for malignancies with low risk of metastasis or death (estimated 5-year overall survival >90%), such as effectively treated early-stage gastrointestinal cancer, carcinoma in situ of the cervix, non-melanoma skin cancer, or localized prostate cancer.
16. Significant comorbid conditions affecting the cardiovascular, respiratory, rheumatological/immunological, hematological, biliary, or pancreatic systems; or history of myocardial infarction, stroke, heart failure, unstable angina, or transient ischemic attack within 6 months prior to screening; or presence of psychiatric disorders.
17. HIV infection.
18. Known allergy or hypersensitivity to rifaximin.
19. Contraindications to MRI, such as incompatible metallic implants, claustrophobia, or body size exceeding scanner capacity.
20. Pregnant or lactating women, women of childbearing potential not using effective contraception, or individuals planning pregnancy.
21. Participation in another investigational drug trial within 3 months prior to screening.
22. Any other condition deemed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The relative change in liver fat content measured by MRI from baseline to 24 weeks. | From enrollment to the end of treatment at 24 weeks
  The relative changes in MRI-measured liver proton density fat fraction (PDFF) at 24 weeks compared to baseline.

SECONDARY OUTCOMES:
The absolute change in liver fat content measured by MRI from baseline to 24 weeks. | From enrollment to the end of treatment at 24 weeks
  Absolute changes in MRI-measured liver proton density fat fraction (PDFF) at 24 weeks compared to baseline.
Proportion of patients achieving ≥30% reduction in liver fat content measured by MRI-PDFF at 24 weeks of treatment compared to baseline | From enrollment to the end of treatment at 24 weeks
  Proportion of patients achieving ≥30% reduction in liver fat content measured by MRI-PDFF at 24 weeks of treatment compared to baseline
The change in liver fat content measured by MRI-PDFF at 12 weeks of treatment | From enrollment to the end of treatment at 12 weeks
  Absolute and relative changes in MRI-measured liver PDFF at 12 weeks compared to baseline.
Proportion of patients achieving ≥30% reduction in liver fat content (PDFF) measured by MRI at 12 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 weeks
  The proportion of patients whose liver fat content (PDFF), assessed via MRI, decreased by ≥30% from baseline after 12 weeks of treatment.
Changes in serum alanine aminotransferase levels after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  Changes in serum ALT levels from baseline after 12 and 24 weeks of treatment
Changes in serum aspartate aminotransferase levels after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  Changes in serum AST levels from baseline after 12 and 24 weeks of treatment
Changes in serum Gamma-Glutamyl Transferase levels after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  Changes in serum GGT levels from baseline after 12 and 24 weeks of treatment
Changes in serum Alkaline Phosphatase levels after 12 and 24 weeks of treatment compared to baseline | From enrollment to the end of treatment at 12 and 24 weeks
  Changes in serum AKP levels from baseline after 12 and 24 weeks of treatment
Change in liver fat content assessed via FibroScan after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  Change in controlled attenuation parameter (CAP) values, measured by FibroScan, from baseline after 12 and 24 weeks of therapy
Changes in fatty liver index (FLI) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  FLI is utilized to assess the severity of hepatic steatosis and is calculated using the following formula: FLI = (e^(0.953 * ln(triglycerides) + 0.139 * BMI + 0.718 * ln(ggt) + 0.053 * waist circumference - 15.745)) / (1 + e^(0.953 * ln(triglycerides) + 0.139 * BMI + 0.718 * ln(ggt) + 0.053 * waist circumference - 15.745)) * 100. Interpretation: A FLI value below 30 can be used to rule out steatosis (sensitivity = 87%; negative likelihood ratio [LR-] = 0.2), while a FLI value equal to or above 60 can be used to rule in hepatic steatosis.
Changes in NAFLD-liver fatty score（NAFLD-LFS）after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  NAFLD-LFS Calculation Formula: NAFLD-LFS = -2.89 + 0.45 × Type 2 Diabetes (yes=2, no=0) + 1.18 × Metabolic Syndrome (yes=1, no=0) + 0.15 × Insulin (mU/L) + 0.04 × AST (U/L) - 0.94 × (AST/ALT Ratio).
  Interpretation of Scores:
  NAFLD-LFS < -1.0: Suggests low liver fat content and a low likelihood of significant steatosis. -1.0 ≤ NAFLD-LFS ≤ 0.5: Intermediate range; further evaluation with additional tests (e.g., imaging or biopsy) is recommended. NAFLD-LFS > 0.5: Indicates high liver fat content and the presence of significant steatosis, requiring clinical intervention.
Changes in AST-to-Platelet Ratio Index (APRI) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  APRI is calculated using the following formula:
  APRI = [ (AST Level (U/L) / AST ULN (Upper Limit of Normal)) / Platelet Count (10⁹/L) ] × 100.
  Interpretation:
  APRI < 0.5: Suggests the absence of significant fibrosis (high negative predictive value). APRI > 2.0: Highly indicative of cirrhosis (high positive predictive value). Intermediate values (0.5 ≤ APRI ≤ 2.0): Further evaluation with additional tests-such as liver elastography, FIB-4 index, or liver biopsy-is recommended for accurate assessment.
Changes in Fibrosis 4 (FIB-4) Score after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 12 and 24 weeks.
  The FIB-4 index is primarily used to stratify the risk of liver fibrosis and is calculated using the following formula: FIB-4= Age (years) × AST (U/L)/ [Platelet Count (10⁹/L)×√ALT(U/L)]. The criteria are categorized as follows: Low Risk (FIB-4 < 1.3) suggests minimal or no fibrosis (F0-F1). Liver biopsy or elastography may be deferred in such cases. Intermediate Risk (1.3 ≤ FIB-4 ≤ 2.67): Further evaluation with additional tests-such as liver elastography, APRI, or liver biopsy-is recommended. Significant fibrosis (F2-F3) may be present, warranting closer monitoring. High Risk (FIB-4 > 2.67): Highly suggestive of advanced fibrosis or cirrhosis (F3-F4). Confirmatory tests like elastography or liver biopsy should be prioritized. This range has a high positive predictive value.
Changes in NAFLD fibrosis score (NFS) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  NFS calculation formula: NFS= [-1.675+0.037×Age (years)+0.094×BMI （kg/m2+1.13×IFG/Diabetes (yes = 1, no = 0) +0.99）× (AST/ALT Ratio)
  +0.013×PLT(×109/L)-0.66×ALB（g/dl）].
  Interpretation Guidelines:
  NFS < -1.455: Low probability of significant fibrosis (F2-F4). NFS > 0.676: High probability of advanced fibrosis (F3-F4). NFS between -1.455 and 0.676: Indeterminate range; further evaluation with additional tests (e.g., elastography or liver biopsy) is recommended.
Changes in FibroScan-AST (FAST) Score after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  The FAST Score is a non-invasive composite index used to assess the likelihood of both significant fibrosis (≥F2) and active steatohepatitis (NASH) in patients withMASLD. It integrates Liver Stiffness Measurement (LSM) obtained via FibroScan® and the serum biomarker AST. FAST Score Calculation Formula: FAST = e^(-1.65 + 1.07 × ln(LSM) + 2.66 × 10^(-8) × AST^3 - 63.3 × AST^(-1) - 0.009 × PLT) / (1 + e^(-1.65 + 1.07 × ln(LSM)
  + 2.66 × 10^(-8) × AST^3 - 63.3 × AST^(-1) - 0.009 × PLT)). Interpretation Guidelines: FAST < 0.35: Low probability of significant fibrosis (≥F2) with active inflammation (NASH). Negative predictive value >90%. Liver biopsy may be avoided. FAST > 0.67: High probability of both significant fibrosis (≥F2) and active inflammation (NASH). Positive predictive value >70%. Further evaluation or intervention is recommended. FAST between 0.35-0.67: Gray zone; comprehensive assessment with additional methods.
Changes in Body Mass Index (BMI) at 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  BMI calculation Formula:
  BMI = Weight (kilograms) ÷ [Height (meters)]²
Changes in Waist circumference (WC) at 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks.
  Waist circumference (WC) is measured 3 cm above the navel.
Changes in visceral adipose tissue (VAT) at 12 and 24 weeks of treatment compared to baseline. [ | From enrollment to the end of treatment at 12 and 24 weeks
  VAT was quantified using 3D Slicer software by manually segmenting regions of interest (ROIs) within the intra-abdominal cavity on MRI images at the level of the third lumbar vertebra (L3).
Changes in abdominal subcutaneous adipose tissue (ASAT) from baseline after 12 and 24 weeks of therapy | From enrollment to the end of treatment at 12 and 24 weeks
  ASAT volume was quantified using 3D Slicer software by manually segmenting regions of interest (ROIs) within the subcutaneous fat compartment on MRI images at the level of the third lumbar vertebra (L3).
Changes in Cholesterol from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks.
  Cholesterol testing should be performed in the morning after an overnight fast.
Changes in triglyceride from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks.
  Triglyceride testing should be performed in the morning after an overnight fast.
Changes in Hemoglobin A1c (HbA1c) from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks.
  Change from baseline in HbA1c absolute concentration (mmol/mol) and percentage of total hemoglobin (%) after 12 and 24 weeks of therapy.
Changes in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  HOMA-IR Calculation Formula: HOMA-IR = [Fasting Insulin (μIU/mL) × Fasting Glucose (mmol/L)] / 22.5. Increase in HOMA-IR suggests worsening insulin resistance. Decrease in HOMA-IR indicates improved insulin sensitivity.
The frequency and severity of treatment-related adverse events (AEs) as assessed by CTCAE 5.0. | From enrollment to the end of treatment at 24 weeks
  The safety assessment involved monitoring changes in symptoms, vital signs, and laboratory parameters during treatment.

OTHER OUTCOMES:
Changes in liver fat content assessed via MRI-PDFF at 12/24 weeks post-treatment. | Through study completion, an average of 2 years
  Longitudinal changes in liver PDFF measured by MRI at 12 and 24 weeks following treatment discontinuation, comparing these time points to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fen Xie, Director, Principal Investigator — Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Locations (1):
- Changzheng Hospital, Naval Medical University, shanghai, China, Shanghai, China